CLINICAL TRIAL: NCT01290497
Title: Pilot, Unicentre, Randomized, Parallel, Controlled Study to Evaluate the Efficacy and Safety of Three Different Intraarticular Dosage Regimens of Adant® in Patients With Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of 3 Different Dosage Regimens of Hyaluronic Acid in Patients With Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tedec-Meiji Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TM-ME3710/403; 2010-021633-31 (EudraCT Number)
Record Dates: First submitted 2011-02-02; First posted 2011-02-07 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hyaluronic acid 5 x 2.5 ml (Active Comparator)
  Interventions: Drug: Hyaluronic acid 5 x 2.5 ml
- Hyaluronic acid 1 X 5 ml (Experimental)
  Interventions: Drug: Hyaluronic acid 1 x 5 ml
- Hyaluronic acid 2 x 5 ml (Experimental)
  Interventions: Drug: Hyaluronic acid 2 x 5 ml

INTERVENTIONS:
Drug: Hyaluronic acid 5 x 2.5 ml — 5 intraarticular administration of Adant® 2.5ml with one week interval between administrations (standard treatment)
  Arms: Hyaluronic acid 5 x 2.5 ml
Drug: Hyaluronic acid 1 x 5 ml — 1 intraarticular administration of Adant® 5ml
  Arms: Hyaluronic acid 1 X 5 ml
Drug: Hyaluronic acid 2 x 5 ml — 2 intraarticular administration of Adant® 5ml with a two-week interval between administrations.
  Arms: Hyaluronic acid 2 x 5 ml

SUMMARY:
The main objective is the comparison of three different dosage regimens of hyaluronic acid in the treatment of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient>45 years of age diagnosed with primary osteoarthritis according to ACR and Kellgren criteria
* Knee pain ≥ 55 mm and ≤90 mm measured by Visual Analogue Scale (VAS) 100 mm
* Ability to understand and follow study procedures
* Written informed consent

Exclusion Criteria:

* Patients with secondary osteoarthritis of the knee according to ACR criteria.
* Severe inflammation of the knee diagnosed by physical examination or a sedimentation speed rate < 40 mm/h and serum rheumatoid factor titre < 1:40
* Patients having previously received surgery, including arthroscopy
* Patients with joint inflammatory disease (spondilitis, systemic rheumatoid arthritis), microcrystalline arthropathies (chondrocalcinosis, gout, fibromyalgia) and significant osteoarthritis symptoms in other joints apart from the knee, and which require pharmacological treatment
* Previous administration of any of the following treatments: hyaluronic acid ia (last year); steroids i.a. or joint lavage (last 3 months), glucosamine sulfate, chondroitin sulfate or diacerein (last 3 months), NSAIDs (last 14 days), any investigational drug (last month) or its administration during this study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The main objective is to evaluate the efficacy of different dosage regimens of intraarticular Hyaluronic Acid 5 ml (Adant®)compared to a standard treatment (2.5ml X 5 i.a) in patients with osteoarthritis of the knee. | 1 year
  Primary endpoint: Pain, Function and patient's assessment according to OARSI 2004 responder criteria.
  Every patient who has received 100% of injections by the end of the study and has fulfilled the follow-up visits will be considered evaluable.
  The percentage of patients in each group who do not complete the study due to lack of efficacy will be evaluated.

SECONDARY OUTCOMES:
To evaluate the safety of the different dosage regimens | 1 year
  Safety endpoints: Recording of adverse events and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Escudero, Principal Investigator
Locations (1):
- Hospital Reina Sofia, Córdoba, Andalusia, Spain